CLINICAL TRIAL: NCT03847181
Title: Safety and Effectiveness of Rivaroxaban and Apixaban Compared to Warfarin in Non-valvular Atrial Fibrillation Patients in the Routine Clinical Practice in the UK
Brief Title: Study to Learn More About the Benefits and Side-effects of Drugs Rivaroxaban and Apixaban Compared to the Drug Warfarin for Stroke Prevention in Patients With Rapid and Irregular Heartbeat Which is Not Due to a Heart-valve Fault (Non-valvular Atrial Fibrillation) in the UK Routine Clinical Practice
Acronym: SiERRA UK
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: 20343; EUPAS28234 (Other: ENCePP)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
Keywords: Oral anticoagulants; Under-dosing; Stroke prevention in atrial fibrillation; Safety; Effectiveness
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; apixaban; Warfarin; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NVAF-patients_1: Adult patients with non-valvular atrial fibrillation (NVAF) and one year health records in the British THIN-database, who have not yet used rivaroxaban, apixaban and warfarin.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- NVAF-patients_2: Adult patients with non-valvular atrial fibrillation (NVAF) and one year health records in the British THIN-database, who have not yet used rivaroxaban, apixaban and warfarin.
  Interventions: Drug: Apixaban (Eliquis)
- NVAF-patients_3: Adult patients with non-valvular atrial fibrillation (NVAF) and one year health records in the British THIN-database, who have not yet used rivaroxaban, apixaban and warfarin.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban at a dose of 15 or 20 mg once daily
  Other Names: Non-Vitamin K Oral Anticoagulant (NOAC)
  Groups: NVAF-patients_1
Drug: Apixaban (Eliquis) — Apixaban at a dose of 2.5 or 5 mg twice daily
  Other Names: Non-Vitamin K Oral Anticoagulant (NOAC)
  Groups: NVAF-patients_2
Drug: Warfarin — Warfarin dose as prescribed by medical practitioner
  Other Names: Vitamin K Antagonist
  Groups: NVAF-patients_3

SUMMARY:
This population-based study will identify patients with rapid and irregular heartbeat which is not due to a fault with the heart valves (non-valvular atrial fibrillation) who initiate rivaroxaban, apixaban or warfarin as treatment for Stroke Prevention in Atrial Fibrillation (SPAF). Purpose of the study is to learn more about the safety and how well the drugs rivaroxaban, apixaban and warfarin work in patients appropriately and inappropriately receiving standard and reduced doses of each drug for reducing the risk of stroke in atrial fibrillation. Real world data from routine general practice stored in the primary care database in the UK, The Health Improvement Network (THIN), will be used for investigation.

DETAILED DESCRIPTION:
Primary objectives are to assess the safety and effectiveness of rivaroxaban, apixaban and warfarin based on the risk of intracranial hemorrhage and hemorrhagic strokes (safety) and ischemic stroke, systemic embolism and myocardial infarction (effectiveness). Secondary objectives comprise the assessment of the mentioned risks in subpopulations of patients with renal impairment or diabetes, mortality rates, and drug utilisation as well as patient characteristics before and after the first intracranial hemorrhage or ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation
* New users of rivaroxaban, apixaban or warfarin
* At least one year enrollment with the general practice (GP)
* One year since first health contact recorded in THIN prior to the first prescription of a study drug

Exclusion Criteria:

* Patients with other recent indications of oral anticoagulant initiation
* Individuals on more than one oral anticoagulant on the start date
* Users of rivaroxaban apart from 15 / 20 mg daily dose
* Users of apixaban apart from 5 / 10 mg daily dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK population sample representative for age, sex and geographic distribution
Sampling Method: Non-Probability Sample
Enrollment: 45164 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Risk of intracranial hemorrhage | Retrospective analysis of data from 2012 to 2017
  Intracranial hemorrhage includes intracerebral hemorrhage, subarachnoid hemorrhage, subdural and epidural hemorrhage.
Risk of ischemic events | Retrospective analysis of data from 2012 to 2017
  Ischemic events include ischaemic stroke / systemic embolism and myocardial infarction.

SECONDARY OUTCOMES:
Risk of intracranial hemorrhage in NVAF-patients with renal impairment | Retrospective analysis of data from 2012 to 2017
  Intracranial hemorrhage includes intracerebral hemorrhage, subarachnoid hemorrhage, subdural and epidural hemorrhage.
Risk of ischemic events in NVAF-patients with renal impairment | Retrospective analysis of data from 2012 to 2017
  Ischemic events include ischaemic stroke / systemic embolism and myocardial infarction.
Risk of intracranial hemorrhage in NVAF-patients with diabetes | Retrospective analysis of data from 2012 to 2017
  Intracranial hemorrhage includes intracerebral hemorrhage, subarachnoid hemorrhage, subdural and epidural hemorrhage.
Risk of ischemic events in NVAF-patients with diabetes | Retrospective analysis of data from 2012 to 2017
  Ischemic events include ischaemic stroke / systemic embolism and myocardial infarction.
All-cause mortality | Retrospective analysis of data from 2012 to 2017
  Rate of deaths from all causes.
Drug utilisation | Retrospective analysis of data from 2012 to 2017
  Drug utilisation comprises a descriptive analysis of characteristics of index prescription, time trends and drug discontinuation.
Drug utilisation after first intracranial hemorrhage or ischemic stroke | Retrospective analysis of data from 2012 to 2017
  Drug utilisation comprises a descriptive analysis of characteristics of index prescription, time trends and drug discontinuation.
Patient characteristics | Retrospective analysis of data from 2012 to 2017
  Patient characteristics comprise a descriptive analysis of baseline characteristics, comorbidities, co-medications and time trends.
Patient characteristics after first intracranial hemorrhage or ischemic stroke | Retrospective analysis of data from 2012 to 2017
  Patient characteristics comprise a descriptive analysis of baseline characteristics, comorbidities, co-medications and time trends.

CONTACTS AND LOCATIONS:
Locations (1):
- Many facilities, Many Sites, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.